CLINICAL TRIAL: NCT05901233
Title: Telerehabilitation With Remotely-Supervised tDCS in Progressive Aphasia
Brief Title: Speech-Language Treatment With Remotely Supervised Transcranial Direct Current Stimulation in Primary Progressive Aphasia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Maya Henry, Associate Professor of Speech, Language and Hearing Sciences, University of Texas at Austin
Allocation: Non-Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00002453
Record Dates: First submitted 2023-05-08; First posted 2023-06-13 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Primary Progressive Aphasia
Keywords: Speech-Language Pathology; Primary Progressive Aphasia; Fronto-Temporal Dementia; Alzheimer's Disease; Neurodegenerative Disease; Logopenic; Semantic; Nonfluent; Logopenic Variant Primary Progressive Aphasia; Semantic Variant Primary Progressive Aphasia; Nonfluent Variant Primary Progressive Aphasia; Semantic Dementia; Speech Entrainment; Script Training; Teletherapy; Transcranial Direct Current Stimulation; Remotely-Supervised Transcranial Direct Current Stimulation; Lexical Retrieval; Noninvasive Brain Stimulation; Telehealth
MeSH Terms: conditions — Aphasia, Primary Progressive; Alzheimer Disease; Neurodegenerative Diseases; Frontotemporal Dementia

STUDY DESIGN:
Intervention Model Description: Participants undergo 4 weeks of video-implemented script training (VISTA) or Lexical Retrieval Training (LRT) with either sham or tDCS, a 2-month washout phase, and then another 4 weeks of LRT or VISTA with the other condition (sham or tDCS). Order will be randomized.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The order of administration for active and sham stimulation phases will be masked for the participant, study partner, study clinician, and primary investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- RS-LRT (Experimental)
  Interventions: Device: Remotely supervised Transcranial Direct Current Stimulation (RS-tDCS); Device: Remotely supervised sham tDCS (RS-sham-tDCS); Behavioral: Lexical Retrieval Training (LRT)
- RS-VISTA (Experimental)
  Interventions: Device: Remotely supervised Transcranial Direct Current Stimulation (RS-tDCS); Device: Remotely supervised sham tDCS (RS-sham-tDCS); Behavioral: Video Implemented Script Training in Aphasia (VISTA)

INTERVENTIONS:
Device: Remotely supervised Transcranial Direct Current Stimulation (RS-tDCS) — tDCS is a type of non-invasive brain stimulation. 1.5 milliamp (mA) of current will be delivered via electrodes in saline-soaked sponges placed on the left side of the head and right upper arm. The stimulation will be delivered for 20 minutes, 5 times weekly, in the participant's home setting while the participant engages in computer-delivered speech-language training. Sessions are monitored by study personnel.
Device: Remotely supervised sham tDCS (RS-sham-tDCS) — tDCS is a type of non-invasive brain stimulation. During sham stimulation 1.5 milliamp (mA) of current will be delivered for a brief period and then turned off. Current will be delivered via electrodes in saline-soaked sponges placed on the left side of the head and right upper arm. Sham will be delivered for 20 minutes, 5 times weekly, in the participant's home setting while the participant engages in computer-delivered speech-language training. Sessions are monitored by study personnel.
Behavioral: Lexical Retrieval Training (LRT) — Participants work on producing spoken and written names of personally relevant target items using a self-cueing hierarchy. Treatment focuses on the use of strategies that capitalize on spared cognitive-linguistic abilities to support word retrieval. The participant completes two (one hour each) teletherapy sessions per week with a clinician plus 30 minutes of additional independent, computer-based practice exercises 3 times per week.
  Arms: RS-LRT
Behavioral: Video Implemented Script Training in Aphasia (VISTA) — Participants work on producing personally relevant scripts of 4-6 sentences in length. Length and complexity of scripts are individually tailored. The participant completes two (one hour each) teletherapy sessions per week with a clinician targeting clear and accurate script production, script memorization, and conversational usage of scripts. The participant completes 30 minutes of independent, computer-based practice 3 times per week, during which they speak in unison with a video/audio model of a healthy speaker clearly articulating the scripts.
  Arms: RS-VISTA

SUMMARY:
Primary progressive aphasia (PPA) is a disorder characterized by gradual decline in speech-language ability caused by underlying neurodegenerative disease. PPA is a devastating condition that can affect adults as young as their 50's, depriving them of the ability to communicate and function in society. Along with Alzheimer's Disease and other Alzheimer's Disease Related Dementias (AD/ADRD), PPA is now identified earlier and with greater precision. Increasingly, patients and families seek options for behavioral and neuromodulatory treatments to address PPA's devastating effects on communication, prolong speech-language skills, and maximize quality of life. Studies have documented the robust benefits of speech-language telerehabilitation methods for persons with PPA, with in-home treatment resulting in immediate and long-term benefits. This investigation aims to further enhance the potency of these treatment approaches by pairing them with tailored neuromodulatory intervention that targets critical brain networks supporting treatment in each clinical subtype of PPA. The study will evaluate the feasibility and preliminary benefit of home-based transcranial direct current stimulation (tDCS) combined with evidence-based speech-language telerehabilitation methods. tDCS will be delivered to patients in their own homes and site of stimulation will be tailored for each clinical subtype of PPA. This project has the potential to enhance clinical management and rehabilitation for individuals with PPA by establishing the benefit of behavioral and neuromodulatory treatment that is neurobiologically-motivated and accessible for patients and families.

ELIGIBILITY:
Because PPA is a rare disease, the study aims to recruit all eligible participants with PPA who are referred to the Aphasia Research and Treatment Lab at the University of Texas (UT) Austin, the UT/Dell Medical School Department of Neurology, and the University of California at San Francisco (UCSF) Memory and Aging Center, as well as individuals with PPA from other clinical and research sites. The study will aim to include males, females, and transgender or non-binary individuals. Great efforts will be made to recruit participants from minority populations, subject to the limitation that participants need to be fluent speakers of English.

Inclusion Criteria:

* Meets diagnostic criteria for PPA
* Meets diagnostic criteria for a specific variant of PPA
* Score of 20 or higher on the Mini-Mental State Examination
* Adequate hearing and vision (with hearing or vision aids, if needed)
* Has a study partner that can co-enroll in the study and attend pre-treatment training as well as continue to be present for weekly teleconference meetings
* Able and willing to undergo MRI brain scan
* Access to high speed internet

Exclusion Criteria:

* Speech and language deficits better accounted for by another neurological disorder
* Does not meet diagnostic criteria for a specific variant of PPA
* Score of less than 20 on the Mini-Mental State Examination
* Does not have a study partner who can co-enroll in the study
* Contraindications for tDCS or MRI scan (History of seizures, head injury, craniotomy, skull surgery or fracture; History of severe or frequent migraines; Metallic implant in head or any metal in head; Pacemaker or cardioverter-defibrillator or any other stimulator; Chronic skin problems; Pregnancy)
* History of stroke, epilepsy, or significant brain injury

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
RS-LRT arm: Change in spoken naming | change from pre-treatment to one month and three months after onset of treatment in each phase (stimulation and sham)
  Change in percent correctly named trained/untrained pictures
RS-VISTA arm: Change in script production accuracy | change from pre-treatment to one month and three months after onset of treatment in each phase (stimulation and sham)
  Change in percent correct, intelligible, scripted words produced for trained/untrained scripts

SECONDARY OUTCOMES:
Change on Communication Confidence Rating Scale for Aphasia | change from pre-treatment to one month and three months after onset of treatment in each phase (stimulation and sham)
  Change on 10-item Likert-type self-rating scale evaluating communication confidence in different settings for persons with aphasia. A higher score indicates greater confidence.
Change on Aphasia Impact Questionnaire | change from pre-treatment to one month and three months after onset of treatment in each phase (stimulation and sham)
  Change on Patient Reported Outcome Measure for persons with aphasia; characterizes activities, participation and emotional state/wellbeing using a 5-point pictorial rating scale. A higher score indicates greater impact of aphasia.
Client Satisfaction Questionnaire | four months after treatment onset
  Likert-type scale measuring patient/client satisfaction with intervention. A higher score indicates greater satisfaction.
Remotely-supervised Transcranial Direct Current Stimulation (RS-tDCS) Survey | four months after onset of treatment
  Likert type scale used to capture participants' perceptions regarding the acceptability and potential demand for remotely-supervised tDCS.
Care Partner Survey | four months after onset of treatment
  Likert-type scale used to characterize care partners' perceptions of the benefits of speech-language treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Maya Henry, PhD, Principal Investigator — University of Texas at Austin
Locations (2):
- United States (2):
  - Memory and Aging Center, University of California, San Francisco, San Francisco, California
  - University of Texas, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Henry ML, Hubbard HI, Grasso SM, Mandelli ML, Wilson SM, Sathishkumar MT, Fridriksson J, Daigle W, Boxer AL, Miller BL, Gorno-Tempini ML. Retraining speech production and fluency in non-fluent/agrammatic primary progressive aphasia. Brain. 2018 Jun 1;141(6):1799-1814. doi: 10.1093/brain/awy101. PMID 29718131
- [Background] Henry ML, Hubbard HI, Grasso SM, Dial HR, Beeson PM, Miller BL, Gorno-Tempini ML. Treatment for Word Retrieval in Semantic and Logopenic Variants of Primary Progressive Aphasia: Immediate and Long-Term Outcomes. J Speech Lang Hear Res. 2019 Aug 15;62(8):2723-2749. doi: 10.1044/2018_JSLHR-L-18-0144. Epub 2019 Aug 7. PMID 31390290
- [Background] Dial HR, Hinshelwood HA, Grasso SM, Hubbard HI, Gorno-Tempini ML, Henry ML. Investigating the utility of teletherapy in individuals with primary progressive aphasia. Clin Interv Aging. 2019 Feb 25;14:453-471. doi: 10.2147/CIA.S178878. eCollection 2019. PMID 30880927
- See also: University of Texas Aphasia Research and Treatment Lab — https://slhs.utexas.edu/research/aphasia-research-treatment-lab
- See also: UCSF Language Neurobiology Lab — https://albalab.ucsf.edu